CLINICAL TRIAL: NCT02211430
Title: Smoking Cessation for Low-Income Pregnant Women
Acronym: ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-832; TURSG-02-227-01-PBP (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2014-05-13; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Pregnancy; Smoking
Keywords: smoking cessation; pregnancy; postpartum; intervention
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioral Counseling (CBC) (Experimental): Cognitive-Behavioral Counseling (CBC) consists of two 45-minute on-site intervention sessions (session 1 and 3), one 15 minute on-site session (session 2), and one 15-minutes phone session (booster session).
  Interventions: Behavioral: Cognitive-Behavioral Counseling (CBC)
- Best Practice (BP) Control (Active Comparator): Best Practice (BP) Control Condition consists of two 10-15 min, on-site intervention sessions (session 1 and 3), one brochure pick-up (session 2), and receipt of a newsletter by mail (booster session).
  Interventions: Behavioral: Best Practice (BC) Control

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Counseling (CBC) — Participants of CBC were educated about the effects of smoking on their personal health and their pregnancy during session 1 (45 minutes counseling), and were encouraged to explore their risk perceptions and emotions, for themselves and their unborn child. During session 2, the 15-minute counseling segment highlighted the cognitive and emotion barriers undermining the participant's motivation to quit and the self-regulatory techniques for resisting personal smoking triggers. Session 3 (45 minutes counseling) involved reviewing smoking status and smoking history over the course of the pregnancy, as well as the effects of smoking on both their health and the health of their infant. Booster session was held by phone for 15 min.
  Arms: Cognitive-Behavioral Counseling (CBC)
Behavioral: Best Practice (BC) Control — For ethical considerations, and consistent with practice guidelines for treating tobacco addiction (Fiore et al., 2000) which mandates that every pregnant smoker be offered smoking cessation treatment, the control group has been designed to be comparable to the current "best practice" guidelines for smoking cessation treatments. This condition, devised from a review of the current literature, will include one brief (5-15 minutes) prenatal individual session (session 1) consisting of smoking cessation education and advice, on-site brochure pick up (session 2), and a second brief postpartum individual session (session 3) followed by receipt of a newsletter (session 4).
  Arms: Best Practice (BP) Control

SUMMARY:
To meet the Healthy People 2010 objective of increasing tobacco abstinence among pregnant women to 90%, new methods for treating nicotine addiction among pregnant women are needed. To this end, we propose to evaluate an innovative cognitive-behavioral smoking cessation intervention for low-income, minority women conducted in the prenatal and postpartum phases. Considering the strong link between tobacco use and cancer risk, the development of effective smoking cessation treatments has important health implications for cancer prevention and control initiatives. The aims to be addressed are:

Aim 1: To compare an enhanced Cognitive-Behavioral Counseling (CBC) smoking cessation intervention with a Best Practice control condition (BP) for reducing smoking rates (i.e., continued abstinence, 7-day point prevalence, and number of cigarettes smoked) in the short- and long-term among pregnant women. It is hypothesized that smokers receiving CBC will show reduced rates of tobacco use, versus those in the BP, over time.

Aim 2: To evaluate the impact of the CBC intervention on the hypothesized mediators of behavior change (i.e., heightened risk perceptions; enhanced self-efficacy and reduced fatalistic beliefs; high pros and low cons of quitting; reduced emotional distress). It is hypothesized that the psychosocial factors will mediate the effect of the CBC intervention on change of smoking behaviors.

DETAILED DESCRIPTION:
Rates of Smoking Among Pregnant and Postpartum Women.

Despite the well-established health risks of prenatal and postpartum smoking, a sizable number of pregnant women and new mothers smoke. About 30% of US women who become pregnant smoke. Only 20-40% of these women spontaneously quit upon learning of their pregnancy. Although an additional 3-16% of pregnant smokers may quit later in pregnancy, the majority continue to smoke throughout, with 15-30% relapsing. Research has also indicated that smoking cessation rates are lower among low-income pregnant women (6-14%) versus more affluent populations. Less educated, lower SES, unemployed women who have a higher addiction to nicotine are at greatest risk for smoking throughout their pregnancy, while pregnant women with higher levels of education and income are more likely to quit. These differential smoking rates result in elevated rates of high-risk pregnancies for low SES and less educated women, vs. higher SES and educated women. While some research has demonstrated moderate success with prenatal smoking cessation interventions, relapse remains a prominent concern. Indeed, more than a quarter of women who quit spontaneously relapse by 6-weeks postpartum, with relapse rates reported as high as 60-80% by 6-months postpartum. The highest relapse rates have been found among women with low income and little education.

Smoking Cessation Interventions for Prenatal and Postpartum Women.

To date, the efficacy of available smoking cessation interventions has been disappointing. The current literature on tobacco control indicates that cognitive-affective factors (including perceived risk, self-efficacy, fatalism, decisional balance, and affect) need to be considered when designing smoking cessation protocols. Yet, the behavioral treatments that have been tested for pregnant smokers focus on the use of self-help guides, basic skills training, and education, neglecting the individual's cognitive-affective profile of barriers. This limitation is paralleled by a similar void in the broader smoking cessation literature. When these characteristics are addressed, they have been considered in isolation, without attention to the full spectrum of cognitive-affective barriers to quitting (i.e., the interventions focus on only 1 barrier such as perceived risk or depression). Not surprisingly, among intervention studies with pregnant women, only 3 produced quit rates above 20%.

Thus, research now needs to build upon these guidelines to develop more potent smoking cessation interventions. The design of our intervention is directly responsive to the call for the development of more creative and powerful behavioral interventions to replace the current best available programs. Guided by the Cognitive-Social Health Information Processing (C-SHIP) model and based on our related behavior change protocols for low-income populations, our approach is tailored to the woman's cognitive-affective profile of barriers to initial, and sustained, uptake of smoking cessation.

Determinants of Smoking Cessation Among Pregnant Women.

The exploration of psychological factors as potential mediators of behavior change appears to be particularly promising. The specific cognitive and affective processes proposed by the C-SHIP model as determinants of the uptake of individual health-protective behaviors (e.g., smoking cessation) include: 1) perceived risk; 2) self-efficacy and fatalistic beliefs; 3) expectancies of consequences (i.e., the pros and cons of cessation); and 4) emotional distress. Over the past decade, a sizable literature has accumulated with respect to the psychological correlates of smoking behavior.

Procedures and Interventions

Women who were between 1-25 weeks gestation were asked to participate in a study aimed at learning about smoking cessation techniques for quitting and relapse prevention. Following recruitment and informed consent, participants were randomly assigned to one of two groups, which varied in intensity: 1) the control group, which provided a brief counseling of educational advice and assistance for quitting during each session or 2) a more intensive theoretically-guided smoking cessation intervention group based on the team's Cognitive-Social Health Information Processing Model (C-SHIP ), which assessed and addressed the participant's distinctive pattern of risk perceptions, expectancies and beliefs, and affective reactions. Through prompts and role-play exercises in the context of in-person counseling, potential barriers to cessation can be triggered in a safe, supportive environment. Baseline and follow-up assessments were conducted at 13-25 weeks gestation, 26-38 weeks gestation, 2-6 weeks postpartum and 20-22 weeks postpartum.

Best Practice (BP) control condition consisted of two on-site 10-15 minutes sessions (session 1 and 3), pick up a smoking cessation guide/brochure (session 2), and receive an educational new letter by mail (booster session). CBC intervention included two 45 minutes on-site counseling sessions session 1 and 3), one 15-minutes on-site counseling session (session 2), and one 15-minutes phone session (booster session).

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant
* Having smoked one puff of a cigarette in the 30 days prior to recruitment (1- 25 weeks post-gestation)
* Being 18 years or older
* Being reachable by a telephone.

Exclusion Criteria:

* An inability to communicate readily in English
* Receiving substance abuse treatment and/or evidence of drug and alcohol abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2002-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Status | prepartum follow-up (26-38 weeks gestation)
  Self-reported quit status will be assessed using continuous abstinence and 7-day point prevalence. Assessment of continuous abstinence consists of interviewing the participant to record their smoking practices on each day from the preceding data point to the current interview date (e.g., duration between the quit date and the end of treatment). In addition, saliva cotinine level will be examined to validate self-report smoking status. Participants with a cotinine level of 10mg or above will be considered smokers. In the case of discrepancies between self-report and biochemical verification from saliva samples, the cotinine level will be used as the criterion.
Smoking Cessation Status | postpartum follow-up (2-6 weeks postpartum)
  Self-reported quit status will be assessed using continuous abstinence and 7-day point prevalence. Assessment of continuous abstinence consists of interviewing the participant to record their smoking practices on each day from the preceding data point to the current interview date (e.g., duration between the quit date and the end of treatment). In addition, saliva cotinine level will be examined to validate self-report smoking status. Participants with a cotinine level of 10mg or above will be considered smokers. In the case of discrepancies between self-report and biochemical verification from saliva samples, the cotinine level will be used as the criterion.
Smoking Cessation Status | 3-month post intervention follow up (20-22 weeks postpartum)
  Self-reported quit status will be assessed using continuous abstinence and 7-day point prevalence. Assessment of continuous abstinence consists of interviewing the participant to record their smoking practices on each day from the preceding data point to the current interview date (e.g., duration between the quit date and the end of treatment). In addition, saliva cotinine level will be examined to validate self-report smoking status. Participants with a cotinine level of 10mg or above will be considered smokers. In the case of discrepancies between self-report and biochemical verification from saliva samples, the cotinine level will be used as the criterion.

SECONDARY OUTCOMES:
Average Number of Cigarettes Smoked Per Day in Past 7 Days | prepartum follow-up (26-38 weeks gestation)
  Participants will be asked to indicate how many cigarettes they smoked per day on average in the past 7 days at baseline and each follow-up.
Average Number of Cigarettes Smoked Per Day in Past 7 Days | postpartum follow-up (2-6 weeks postpartum)
  Participants will be asked to indicate how many cigarettes they smoked per day on average in the past 7 days at baseline and each follow-up.
Average Number of Cigarettes Smoked Per Day in Past 7 Days | 3-month post intervention follow up (20-22 weeks postpartum)
  Participants will be asked to indicate how many cigarettes they smoked per day on average in the past 7 days at baseline and each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Miller, Ph.D., Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] DiClemente CC, Dolan-Mullen P, Windsor RA. The process of pregnancy smoking cessation: implications for interventions. Tob Control. 2000;9 Suppl 3(Suppl 3):III16-21. doi: 10.1136/tc.9.suppl_3.iii16. PMID 10982900
- [Background] Engstrom, P., Clapper, M., Schnoll, R., & Orleans, C.T. (2000). Prevention of tobacco-related cancers. Baltimore, MD: Williams and Wilkins Publishing.
- [Background] Miller, S.M. (2000). Tobacco-related cancers can be prevented and controlled. Primary Care & Cancer, 20(6), 8-9.
- [Background] Miller, S.M., & Diefenbach, M. (1998). C-SHIP: A cognitive-social health information processing approach to cancer. In D. Krantz (Ed.), Perspectives in behavioral medicine. New Jersey: Lawrence Erlbaum.
- [Background] Miller SM, Rodoletz M, Mangan CE, Schroeder CM, Sedlacek TV. Applications of the monitoring process model to coping with severe long-term medical threats. Health Psychol. 1996 May;15(3):216-25. doi: 10.1037//0278-6133.15.3.216. PMID 8698036
- [Background] Miller SM, Shoda Y, Hurley K. Applying cognitive-social theory to health-protective behavior: breast self-examination in cancer screening. Psychol Bull. 1996 Jan;119(1):70-94. doi: 10.1037/0033-2909.119.1.70. PMID 8559860
- [Background] Miller, S. M., & Schnoll, R.A. (2000). Coping with stress: examples from the cancer context. In J. M. M. Lewis (Ed.), Handbook of Emotions. NY, NY: Plenum Press.
- [Background] Orleans CT, Boyd NR, Bingler R, Sutton C, Fairclough D, Heller D, McClatchey M, Ward JA, Graves C, Fleisher L, Baum S. A self-help intervention for African American smokers: tailoring cancer information service counseling for a special population. Prev Med. 1998 Sep-Oct;27(5 Pt 2):S61-70. doi: 10.1006/pmed.1998.0400. PMID 9808825
- [Background] Zapka JG, Pbert L, Stoddard AM, Ockene JK, Goins KV, Bonollo D. Smoking cessation counseling with pregnant and postpartum women: a survey of community health center providers. Am J Public Health. 2000 Jan;90(1):78-84. doi: 10.2105/ajph.90.1.78. PMID 10630141
- [Background] Aakko E, Piasecki TM, Remington P, Fiore MC. Smoking cessation services offered by health insurance plans for Wisconsin state employees. WMJ. 1999 Jan-Feb;98(1):14-8. PMID 10050148
- [Background] Adams MM, Brogan DJ, Kendrick JS, Shulman HB, Zahniser SC, Bruce FC. Smoking, pregnancy, and source of prenatal care: results from the Pregnancy Risk Assessment Monitoring System. The Pregnancy Risk Assessment Monitoring System Working Group. Obstet Gynecol. 1992 Nov;80(5):738-44. PMID 1407908
- [Background] Botvin GJ, Epstein JA, Botvin EM. Adolescent cigarette smoking: prevalence, causes, and intervention approaches. Adolesc Med. 1998 Jun;9(2):299-313, vi. PMID 10961237
- [Background] Dolan-Mullen P, Ramirez G, Groff JY. A meta-analysis of randomized trials of prenatal smoking cessation interventions. Am J Obstet Gynecol. 1994 Nov;171(5):1328-34. doi: 10.1016/0002-9378(94)90156-2. PMID 7977542
- [Background] Ershoff DH, Quinn VP, Mullen PD. Relapse prevention among women who stop smoking early in pregnancy: a randomized clinical trial of a self-help intervention. Am J Prev Med. 1995 May-Jun;11(3):178-84. PMID 7662397
- [Background] Fingerhut LA, Kleinman JC, Kendrick JS. Smoking before, during, and after pregnancy. Am J Public Health. 1990 May;80(5):541-4. doi: 10.2105/ajph.80.5.541. PMID 2327529
- [Background] Fiore, M., Bailey, W., Cohen, S., Dorfman, S., Goldstein, M., Gritz, E., Heyman, R., Jaen, C., Kottke, T., Lando, H., Mecklenburg, R., Dolan-Mullen, P., Nett, L., Robinson, L., Stitzer, M., Tommasello, A., Villejo, L., & Wewers, M. (2000). Treating tobacco use and dependance. Clinical Practic Guideline. Rockville, MD: U.S. Department of Health and Human Services. Public Health Service.
- [Background] Gielen AC, Windsor R, Faden RR, O'Campo P, Repke J, Davis M. Evaluation of a smoking cessation intervention for pregnant women in an urban prenatal clinic. Health Educ Res. 1997 Jun;12(2):247-54. doi: 10.1093/her/12.2.247. PMID 10168576
- [Background] Hartmann KE, Thorp JM Jr, Pahel-Short L, Koch MA. A randomized controlled trial of smoking cessation intervention in pregnancy in an academic clinic. Obstet Gynecol. 1996 Apr;87(4):621-6. doi: 10.1016/0029-7844(95)00492-0. PMID 8602320
- [Background] Hill HA, Schoenbach VJ, Kleinbaum DG, Strecher VJ, Orleans CT, Gebski VJ, Kaplan BH. A longitudinal analysis of predictors of quitting smoking among participants in a self-help intervention trial. Addict Behav. 1994 Mar-Apr;19(2):159-73. doi: 10.1016/0306-4603(94)90040-x. PMID 8036963
- [Background] Kendrick JS, Zahniser SC, Miller N, Salas N, Stine J, Gargiullo PM, Floyd RL, Spierto FW, Sexton M, Metzger RW, et al. Integrating smoking cessation into routine public prenatal care: the Smoking Cessation in Pregnancy project. Am J Public Health. 1995 Feb;85(2):217-22. doi: 10.2105/ajph.85.2.217. PMID 7856781
- [Background] Kowalski SD. Self-esteem and self-efficacy as predictors of success in smoking cessation. J Holist Nurs. 1997 Jun;15(2):128-42. doi: 10.1177/089801019701500205. PMID 9165803
- [Background] Lando HA, Rolnick S, Klevan D, Roski J, Cherney L, Lauger G. Telephone support as an adjunct to transdermal nicotine in smoking cessation. Am J Public Health. 1997 Oct;87(10):1670-4. doi: 10.2105/ajph.87.10.1670. PMID 9357351
- [Background] Lillington L, Royce J, Novak D, Ruvalcaba M, Chlebowski R. Evaluation of a smoking cessation program for pregnant minority women. Cancer Pract. 1995 May-Jun;3(3):157-63. PMID 7599672
- [Background] Matheny KB, Weatherman KE. Predictors of smoking cessation and maintenance. J Clin Psychol. 1998 Feb;54(2):223-35. doi: 10.1002/(sici)1097-4679(199802)54:23.0.co;2-l. PMID 9467767
- [Background] Mayer JP, Hawkins B, Todd R. A randomized evaluation of smoking cessation interventions for pregnant women at a WIC clinic. Am J Public Health. 1990 Jan;80(1):76-8. doi: 10.2105/ajph.80.1.76. PMID 2293809
- [Background] McBride CM, Curry SJ, Lando HA, Pirie PL, Grothaus LC, Nelson JC. Prevention of relapse in women who quit smoking during pregnancy. Am J Public Health. 1999 May;89(5):706-11. doi: 10.2105/ajph.89.5.706. PMID 10224982
- [Background] Mullen PD, Richardson MA, Quinn VP, Ershoff DH. Postpartum return to smoking: who is at risk and when. Am J Health Promot. 1997 May-Jun;11(5):323-30. doi: 10.4278/0890-1171-11.5.323. PMID 10167366
- [Background] O'Connor AM, Davies BL, Dulberg CS, Buhler PL, Nadon C, McBride BH, Benzie RJ. Effectiveness of a pregnancy smoking cessation program. J Obstet Gynecol Neonatal Nurs. 1992 Sep-Oct;21(5):385-92. doi: 10.1111/j.1552-6909.1992.tb01755.x. PMID 1403224
- [Background] Secker-Walker RH, Solomon LJ, Flynn BS, Skelly JM, Lepage SS, Goodwin GD, Mead PB. Individualized smoking cessation counseling during prenatal and early postnatal care. Am J Obstet Gynecol. 1994 Nov;171(5):1347-55. doi: 10.1016/0002-9378(94)90159-7. PMID 7977545
- [Background] Valbo, A., & Schioldborg, P. (1994). Smoking cessation in pregnancy: the effects of self-help manuals. Journal of Maternal Fetal Investigation, 4, 167-170.
- [Background] Valbo A, Nylander G. Smoking cessation in pregnancy. Intervention among heavy smokers. Acta Obstet Gynecol Scand. 1994 Mar;73(3):215-9. doi: 10.3109/00016349409023442. PMID 8122501
- [Background] Walsh RA, Redman S, Brinsmead MW, Byrne JM, Melmeth A. A smoking cessation program at a public antenatal clinic. Am J Public Health. 1997 Jul;87(7):1201-4. doi: 10.2105/ajph.87.7.1201. PMID 9240113
- [Background] Windsor RA, Lowe JB, Perkins LL, Smith-Yoder D, Artz L, Crawford M, Amburgy K, Boyd NR Jr. Health education for pregnant smokers: its behavioral impact and cost benefit. Am J Public Health. 1993 Feb;83(2):201-6. doi: 10.2105/ajph.83.2.201. PMID 8427323